CLINICAL TRIAL: NCT03216694
Title: The Association Between Preoperative Cardiopulmonary Exercise Test Variables and Short-term Postoperative Morbidity Following Oesophagectomy: a Hospital-based Cohort Study
Brief Title: The Association Between Preoperative CPEX and Postoperative Morbidity Following Oesophagectomy
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 222793
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise testing — Aerobic fitness measured using a cycle ergometer and metabolic cart

SUMMARY:
A retrospective hospital-based cohort study of the association between preoperative cardiopulmonary exercise test (CPEX) variables and short-term postoperative morbidity following oesophagectomy.

DETAILED DESCRIPTION:
The aim of this study is to examine the correlations between preoperative CPEX variables (VO2max and Anaerobic Threshold) and 30 day postoperative all cause morbidity in a sample large enough to allow (should significant associations exist) calculation of a threshold value. Secondary aims are to examine associations between the VO2max, AT and cardiopulmonary, non-cardiopulmonary complications as well as specific complications (atrial fibrillation, pneumonia, and anastomotic leak) as well as 30 and 90 day mortality.

ELIGIBILITY:
Inclusion Criteria:

i. male and female ii. underwent an oesophagectomy iii. completed a pre-operative CPEX test

Exclusion Criteria:

i. patients that were unable to complete a full CPEX test ii. emergency or palliative surgery iii. pharyngolaryngo-oesophagectomy iv. oesophagectomy and gastrectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent oeosphagectomy at the Norfolk and Norwich Hospital between September 2011 to March 2017
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
All cause postoperative morbidity | 30 days
  Classified using Esophageal Complications Consensus Group (ECCG) definitions [1] and graded using Clavien-Dindo severity classification [2].

SECONDARY OUTCOMES:
Cardiopulmonary complications | 30 days
  Classified using ECCG definitions and graded using Clavien-Dindo severity classification.
Non-cardiopulmonary complications | 30 days
  Classified using ECCG definitions and graded using Clavien-Dindo severity classification.
Mortality | 30 days
  All cause mortality.
Mortality | 90 days
  All cause mortality.
Pneumonia | 30 days
  Classified using ECCG definitions and graded using Clavien-Dindo severity classification.
Atrial fibrillation | 30 days
  Classified using ECCG definitions and graded using Clavien-Dindo severity classification.
Anastomotic leak | 30 days
  Classified using ECCG definitions and graded using Clavien-Dindo severity classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: [1] — https://www.ncbi.nlm.nih.gov/pubmed/25607756
- See also: [2] — https://www.ncbi.nlm.nih.gov/pubmed/15273542